CLINICAL TRIAL: NCT04646447
Title: Tolerability and Efficacy of L-Serine in Patients With GRIN-related Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIC-29-20
Record Dates: First submitted 2020-09-28; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: GRIN Related Disorders
MeSH Terms: interventions — Serine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- L-serine treatment (Experimental): All patients will receive the same L-serine dose treatment over 12 months. Arm: Experimental: L-Serine 250 mg / kg / day during the first two weeks. From week 3 to 52, 500 mg / kg / day. L-serine orally administered, divided into three doses a day.
  Interventions: Dietary Supplement: L-serine

INTERVENTIONS:
Dietary Supplement: L-serine — L-Serine Arm L-serine is considered as GRAS (generally recognized as safe) by the FDA and has been approved as a normal food additive under CFR172.320.
  All patients will receive the same L-serine dose treatment over 12 months. Arm: Experimental: L-Serine 250 mg / kg / day during the first two weeks. From week 3 to 52, 500 mg / kg / day. L-serine orally administered, divided into three doses a day.
  The L-Serine will be manufactured, packaged, labeled and/or distributed by NUTRICIA or delegated contractors. It will be presented in a powdered form of 100 gr of the amino acid L-serine. For oral use.
  Sufficient L-serine will be dispensed at home considering the dose according the weight of the patient.

SUMMARY:
GRIN-related disorders encompass a new group of Inborn Errors of Metabolism according to the recent nosology published by Ferreira et al (Genet Med, 2019).

These rare conditions represent a subtype of paediatric encephalopathies leading to intellectual disability, hypotonia, communication deficits and motor impairment (Orphanet entries: 178469, 289266, 101685, for GRIN1, GRIN2A and GRIN2B, respectively).

Mutations leading to glutamatergic hypotransmission can be potentially treated with L-Serine leading to significant clinical benefits in patients according to a pilot study published by our group (Soto et al, 2019).

In our study, the investigators will include about 20 spanish patients older than 2 years of age, harbouring GRIN variants functionally anotated as loss-of-function pathogenic variants. The investigators will evaluate dose tolerability, efficacy of the treatment according to neurocognitive and motor scales, as well as the effects of L-serine in microbiome composition.

DETAILED DESCRIPTION:
GRIN-related disorders, a novel group of IEM (inborn errors of metabolism): Mutations on GRIN genes, encoding for the N-methyl-D-Aspartate receptor (NMDAR) subunits, have been recently associated with autosomic dominant GRIN-related disorders (Lemke et al., 2016; Platzer et al., 2017; XiangWei et al., 2018; Strehlow et al., 2019). These rare conditions represent a subtype of paediatric encephalopathies leading to intellectual disability, hypotonia, communication deficits and motor impairment (Orphanet entries: 178469, 289266, 101685, for GRIN1, GRIN2A and GRIN2B, respectively).

There are about 200 patients affected with these diseases in Europe according to a data collection study conducted by the patients' families and presented at the first European meeting of GRIN disorders in October 2018 (Barcelona, Hospital Sant Joan de Déu).

Along the last years, our research efforts were focused to delineate the pathophysiology and personalized therapies for these diseases that are now considered as a new category of IEM. In particular, the recent nosology of inherited metabolic disorders (Ferreira et al, 2018) classifies GRIN-related disorders in the category: "DISORDERS OF NITROGEN CONTAINING COMPOUNDS", and the subgroup: "20. Disorders of glutamate metabolism":

GRIN1 (OMIM138249): Ionotropic glutamate receptor NMDA type subunit 1 dysregulation (AD, AR): Autosomal dominant mental retardation type 8; neurodevelopmental disorder with or without hyperkinetic movements and seizures. GRIN2A (OMIM138253): Ionotropic glutamate receptor NMDA type subunit 2A dysregulation (AD): Non related to human disease so far. GRIN2B (OMIM138252): Inotropic glutamate receptor NMDA type subunit 2B dysregulation (AD): Early infantile epileptic encephalopathy type 27; autosomal dominant mental retardation type 6. GRIN2D (OMIM602717): Ionotropic glutamate receptor NMDA type subunit 2D superactivity (AD): Early infantile epileptic encephalopathy type 46.

Indeed, in a proof-of-concept, the investigators have determined that a GRIN2B loss-of-function variant can be rescued in vitro, by means of elevated doses of D-serine (NMDAR coagonist) administration. More importantly, the investigators showed that L-serine (the D-serine natural precursor) dietary supplement was associated with a significant improvement of motor and communication skills of the patient harbouring GRIN2B hypofunctional variant (Soto et al., 2019).

Serine enantiomers: cognitive enhancement and potential use in GRIN-related disorders L-serine (C3H7NO3; 105.09 g/mol; synonym (S)-2-amino-3-hydroxypropanoic acid) is a naturally-occurring dietary amino acid. It is abundant in soy products, some edible seaweeds, sweet potatoes, eggs, and meat. Since some L-serine is produced by astrocytes in the brain, it is considered a non-essential amino acid. L-serine is directly involved in the biosynthesis of purines, pyrimidines, and other amino acids. Serine residues are found in most proteins and within proteins function as a site for phosphorylation.

L-serine is considered as GRAS (generally recognized as safe) by the FDA and has been approved as a normal food additive under CFR172.320. It is widely sold as a dietary supplement. A randomized trial of L-serine in 18 patients with hereditary sensory and autonomic neuropathy type 1 has been published (ClinicalTrials.gov identifier NCT01733407). High-dose oral L-serine supplementation (400 mg/kg/day) appears safe in patients with HSAN1 and is potentially effective at slowing disease progression.The authors did not report adverse effects at doses of 400mg/kg/day (Eichler et al) Further, L-serine dietary supplement has been used in Paediatrics at doses of 400 to 600 mg/kg/day since several decades ago for the treatment of a group of inherited metabolic disorders, namely: 3-phosphoglycerate dehydrogenase deficiency, phosphoserine aminotransferase deficiency and phosphoserine phosphatase deficiency, with no reported adverse effects. In patients with 3-phosphoglycerate dehydrogenase deficiency, neither 100 nor 200 mg/kg per day had any effects on the patients' symptoms or on CSF serine and glycine concentrations (de Koning et al 1998). Only with L-serine 500 mg/kg per day was a reduction in seizure activity noted and an increase in serine CSF concentrations observed (Koning 2006).

D-serine, the natural coagonist of the NMDA receptor, results from the racemisation of L-serine in brain, and its biosynthetic alteration can lead to neuronal dysfunction (van de Crabben et al., 2013). In addition to its homeostatic role in neuronal function, the beneficial effect of D-serine supplement has been recently shown in healthy individuals (Levin et al., 2015). Heresco-Levy's group showed the procognitive effects of D-serine throughout NMDA receptor function. D-serine deficits have been associated with aging in rats, with a functional rescue observed following D-serine administration (Turpin et al., 2011; Billard, 2015).

Additionally, L-serine biosynthesis defects (de Koning, 2006) cause neurological phenotypes (psychomotor retardation, microcephaly, seizures) that can be safely treated by L-serine.

Moreover, and as already mentioned, our group has recently described the beneficial effect of a chronic L-serine dietary (500 mg/kg/per day) supplement in a 5 years GRIN2B patient (Soto et al., 2019). The patient has shown notable improvements in motor and cognitive performance and communication after 11 and 17 months of L-serine dietary supplementation. These data suggest that L-serine supplementation might ameliorate GRIN2B-related severe encephalopathy and other neurological conditions caused by glutamatergic signaling deficiency.

Besides this direct effect, D-serine can prevent behavioral abnormalities in adult mice challenged by maternal immune activation (Fujita et al., 2016), and induces hippocampal neurogenesis (Sultan et al., 2015).

These evidences indicate that 500 mg/kg/per day is a safe and effective dose, that could be used in patients with GRIN related disorders.

HYPOTHESIS Overall, these evidences indicate that, independently on the molecular aetiology, NMDAR activity potentiation throughout L-serine dietary supplement can ameliorate glutamatergic function and improve the life quality of children suffering from GRIN-related disorders, a novel IEM. Dietary supplement of L-serine results on increased D-serine plasma levels and potentiates NMDA receptors leading to NMDA receptors functionality increase and hypofunctionality rescue, as shown in a pilot study (Soto et al., 2019).

AIM The purpose of this study is to determine L-Serine dietary supplement efficacy for the treatment of patients with GRIN-related disorders caused by the presence of GRIN genetic variants leading to hypofunctional (loss-of-function) NMDA receptors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of encephalopathy associated with genetic GRIN variant pathogenic or likely pathogenic, causing a loss-of-function
* Parent(s)/legal representative give written informed consent for participation in the trial; patient assent (if possessing adequate understanding, in the investigator's)
* Patient & caregiver are willing and able (in the investigator's opinion) to comply with all trial requirements (including the completion of all caregiver assessments by the same caregiver throughout the trial).

Exclusion Criteria:

* Diagnosis of encephalopathy with absence of genetic GRIN variant pathogenic or likely pathogenic.
* Currently using or has used within the 30 days prior to screening L-Serine supplement
* Patient has been previously randomized into this trial

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with any adverse event | up to 12 months
  Dose tolerability is based on subject interviews and scheduled assessment evaluating the presence or absence of adverse events.
  The presence of adverse events will be collected according the doses of L-serine: 250 mg / kg / day and 500 mg / kg / day.
  Pre-existing conditions (present before intake of study nutreceutical) or pretreatment AEs (onset before intake of study nutraceutical) are considered concomitant diseases and should not be recorded as AEs but should be recorded on the concomitant diseases eCRF page. However, if the subject experiences a worsening, increased frequency, or complication of such a concomitant disease, the worsening, increased frequency, or complication should be recorded as an AE.
Change in mental age with Vineland Adaptive Behavior Scales (VABS) (Vineland-3) | Baseline (approximately 3 months prior to intervention), 0 months (start treatment) and 3, 6 and 12 months post intervention
  Exploring the following domains: Communication, Daily Living Skills, Socialization and motor Skills (gross and fine) Once obtained the mental age equivalent, the neuropsychologist test or battery to assess the neurodevelopment will be selected
Change in bayley Scales of Infant and Toddler Development (BSID) | Baseline (approximately 3 months prior to intervention), 0 months (start treatment) and 3, 6 and 12 months post intervention
  The Bayley Scales of Infant and Toddler Development (BSID-III) are a set of standardized rating scales, which enable us to assess the cognition, receptive language, expressive language, fine motor and gross motor of children between 1 and 42 months. The Cognitive battery, which consists on the evaluation of the following items: visual perception, attention, memory, objects manipulation and exploration, communication skills and verbal comprehension.
  Bayley III has a raw score, scale score, composite score, and growth percentile score. All of these scores will be given in the study. A higher score means improvement is better.
  The high score for cognition is 91, 48 for receptive language, 49 for expressive language, 66 for fine motor and 72 for gross motor evaluation.
Efficiency of the treatment measured by change in the cognitive assessment (Wechsler Intelligence Scale. | Baseline (approximately 3 months prior to intervention), 0 months (start treatment) and 3, 6 and 12 months post intervention
  If the mental age is more than 42 months will be considering the followings neuropsychologist test: Specific test will be chosen according the age of the children.
  1. The Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV): Age range: 2 years 6 months to 7 years 7 months. An index score can range from 40 to 160. A higher score means improvement is better.
  2. The Wechsler Intelligence Scale for Children (WISC V): Age range: Children aged 6:0-16:11. It has 5 composite scores and a Full-Scale Intelligence Quotient (FSIQ) is generated based on seven subtests. The primary index scores range from 45 to 155; the FSIQ ranges from 40 to 160. A higher score means improvement is better.
  3. The Wechsler Adult Intelligence Scale (WAIS-IV): Age range: 16 years to 90 years, 11 months. The test has 15 subtests, 10 of which are core subtests that are usually used to measure the four index scores and the FSIQ. A higher score means improvement is better.
Change in the Achenbach System of Empirically Based Assessment (ASEBA) System of Empirically Based Assessment (ASEBA)+ | Baseline (approximately 3 months prior to intervention), 0 months (start treatment) and 3, 6 and 12 months post intervention
  The Achenbach System of Empirically Based Assessment (ASEBA) for parents and teachers offers a comprehensive approach to assessing adaptive and maladaptive functioning
Change in Gross Motor Function Measure-88 | -3 months, 0 months (start treatment), 3 months, 6 months, 12 months
  Items span the spectrum of gross motor activities in five dimensions.
  A: Lying and Rolling, B: Sitting C: Crawling and Kneeling, D: Standing, and E: Walking, Running and Jumping.
Change in Social Communication Questionnaire (SCQ) | Baseline (approximately 3 months prior to intervention), 0 months (start treatment) and 3, 6 and 12 months post intervention
  Evaluates communication skills and social functioning in children who may have autism or autism spectrum disorders and The SCQ is a 40-item survey where each question is a 'yes' or 'no' answer. The total possible range of scores is 0-39 (verbal children) or 0-33 (non-verbal children) with higher scores indicative of greater frequency of symptoms. They are completed by parents or other primary caregiver.
Change in the Sleep Disturbance Scale for Children (SDSC) | Baseline (approximately 3 months prior to intervention), 0 months (start treatment) and 3, 6 and 12 months post intervention
  The Sleep Disturbance Scale for Children (SDSC) is a 27-item inventory rated on a 5 point Likert-type scale. 0 = least severe and 5 = most severe
  The instrument's purpose is to categorize sleep disorders in children. As well as giving an overall score the instrument uses five subdomains: disorders of initiating and maintaining sleep, sleep breathing disorders, disorders of arousal, sleep-wake transition disorders, disorders of excessive somnolence, and sleep hyperhidrosis.

SECONDARY OUTCOMES:
Microbiota composition | [ Time Frame: 12 months ]
  Metagenome analysis of the gastrointestinal tract of GRIN-related disorders individuals

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR